CLINICAL TRIAL: NCT04215159
Title: Prospective Phase II Study to Investigate the Efficacy and Safety of Trastuzumab Biosimilar (Samfenet®) Plus Treatment of Physician's Choice (TPC) in Patients With HER2-positive Unresectable Locally Advanced or Metastatic Solid Tumor
Brief Title: Trastuzumab Biosimilar (Samfenet®) Plus Treatment of Physician's Choice (TPC) in Patients With HER2-positive Solid Tumor
Acronym: BIOs-Her
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jin-Hee Ahn (Other)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jin-Hee Ahn, Clinical Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0989
Record Dates: First submitted 2019-09-24; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: HER-2 Protein Overexpression; HER-2 Gene Amplification
Keywords: HER-2 Protein Overexpression; HER-2 Gene Amplification; HER2 targeted-treatment; Trastuzumab biosimilar; samfenet
MeSH Terms: interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Samfenet and Treatment of physician's choice (Experimental): * Samfenet : 1st cycle 8 mg/kg by IV infusion over 90 mins, from 2nd cycle 6mg/kg by IV infusion over 30 mins. every 3weeks.
  * Treatment of physician's choice (Gemcitabine or Irinotecan)
    1. Gemcitabine : 1000 mg/m2 by IV infusion over 30 minutes on Day 1, Day 8. every 3weeks.
    2. Irinotecan : 100 mg/m2 by IV infusion over 90 minutes on Day 1, Day 8. every 3weeks.
  Interventions: Drug: Trastuzumab biosimilar; Drug: Gemcitabine Hydrochloride; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Trastuzumab biosimilar — 1st cycle 8 mg/kg by IV infusion over 90 mins, from 2nd cycle 6mg/kg by IV infusion over 30 mins. every 3weeks.
  Other Names: Samfenet
Drug: Gemcitabine Hydrochloride — 1000 mg/m2 by IV infusion over 30 minutes on Day 1, Day 8. every 3weeks.
  Other Names: Gemtan
Drug: Irinotecan Hydrochloride — 100 mg/m2 by IV infusion over 90 minutes on Day 1, Day 8. every 3weeks.
  Other Names: Calmtop

SUMMARY:
HER2 signaling pathway abnormalities or HER2 overexpression can be seen in various types of solid tumors apart from breast cancer or hepatic cancer. In this regardHER2 targeting therapy has been proven to be effective in colorectal cancer, gallbladder cancer, and salivary gland tumors. Although HER2 targeted-treatment Trastuzumab biosimilar is clinically being used after gaining official permission recently, clinical data for this use is still lacking, especially regarding experiences of combination with various cytotoxic chemotherapy agents.

Notably, techniques to separate and extract a small sized ciculating tumor DNA (ctDNA) in patient's blood originated from a tumor is being developed and improved along with introduction of Next-generation sequencing (NGS) technique enabling a comprehensive genetic testing.

The aim of this study is to evaluate the efficacy and safety of Trastuzumab biosimiler and to investigate the association between ctDNA and clinical outcomes such as disease response, progression-free survival, and overall survival.

DETAILED DESCRIPTION:
Samfenet is a biosimilar of trastuzumab and received marketing approval based on the results of efficacy equivalence to trastuzumab. This study is a phase 2 study to investigate the efficacy of Samfenet in combination with cytotoxic agents in patients with HER2-positive solid tumors.

A total of 42 patients will be enrolled. Treatment will be continues until disease progression, unacceptable toxicity or patient withdrawal. Tumor evaluation will be performed at every 8 weeks during treatment, and then at every 12 weeks thereafter end of study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2 -overexpression (HER2 overexpression defined as 3+ positive by immunohistochemistry, positive by fluorescence in situ hybridization (FISH), or confirmation of HER2 amplification). However hepatic cancer and breast cancer are exclude as HER2 targeted treatment is already a standard treatment for these tumor types.
* Patients who have progressed after at least one standard treatment or unable to continue standard treatment due to adverse events.
* Patients confirmed as metastatic or unresectable cancer by imaging test
* At least one measurable lesion that can be accurately assessed by imaging according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at trial entry
* Adequate organ function (bone marrow, liver, kidney function) A. ANC ≥ 1000/mL B.Platelets ≥ 75,000/uL C.Hemoglobin >8.0 g/dL D.Total bilirubin ≤ 2.0x ULN E.AST and ALT < 5.0 x ULN F.Alkaline phosphatase <2.5x ULN GCreatinine ≤ 2.0x ULN or CCr >30 ml/min
* Estimated life expectancy of more than 3 months
* Left ventricular ejection fraction of at least ≥ 50% at trial entry
* Age ≥19 years who have signed an informed consent approved by Institutional Review Board of Organization

Exclusion Criteria:

* Either woman of pregnancy or breast-feeding woman who is positive for hCG
* Symptomatic or unstable metastases to central nervous system (exceptions : properly treated brain metastasis with no evidence of progression on CT or MRI scan compared with prior examination and without requirement for steroid therapy for relief of symptom. Treatment of an anticonvulsant of stable dose for more than 4 months is permitted taken.
* Evidence of viral, bacterial, or fungal infection including active hepatitis C and D or HIV infection.
* Underwent major surgery of have not fully recovered from certain procedures within 4 months prior to taking the investigational product
* History of malignant disease within 3 years prior to taking the investigational product (exceptions: treated carcinoma in situ of cervix, differentiated thyroid cancer without lymph node metastasis, and skin cancer other than melanoma).
* Interval of QTc > 480 msec (in terms of average measurement of EKG 3 times), oneself or family known to be long or short QT, brugada syndrome or other known QTc prolongation history or Torsade de Pointes.
* Following symptoms or disease within 6 months prior to taking the investigational product: myocardiac infarction, NCI CTCAE v 5.0 Grade ≤2 severe/unstable angina, continuous arrhythmia, atrial fibrillation, bypass surgery of coronary or peripheral arteries, symptomatic heart failure, cerebrovascular events including transient ischemic attack, or symptomatic pulmonary embolism.
* History of symptomatic interstitial lung disease
* Hypersensitivity reaction to Trastuzumab, Gemcitabine, Irinotecan or components of these agents
* Patients with diarrhea, intestinal paralysis, intestinal obstruction, massive ascites, or pleural effusion
* Other psychiatric problems, suicidal attempt, abnormal test results that can affect the administration of the investigational product or participation of clinical trial or that can impact the results of the clinical trial, and any other reason that investigator acknowledge as unsuitable factor for participating the clinical trial.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-12-30 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 8 weeks
  Best response according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  PFS is defined as the time from the first dose of trial treatment to the date of disease progression or death due to any cause, whichever occurs first.
overall survival (OS) | 3 years
  OS is defined as the time from the first dose of trial treatment to the death of all causes or the last follow-up.
Safety profile: NCI-CTCAE | 3 years
  Adverse events graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03

IPD SHARING:
Plan to Share IPD: No